CLINICAL TRIAL: NCT07100314
Title: Impact of Preoperative Toxicological Screening on Perioperative Anesthetic Management and Short-Term Outcomes Following Metabolic Bariatric Surgery: An Observational Study.
Brief Title: Preoperative Toxicological Screening on Perioperative Anesthetic Management
Status: Completed | Type: Observational
Sponsor: General Committee of Teaching Hospitals and Institutes, Egypt (Other Government)
Responsible Party: Principal Investigator, Mohamed Hany Ashour, Professor of General surgery, General Committee of Teaching Hospitals and Institutes, Egypt
Other Study IDs: Preoperative Toxicology
Record Dates: First submitted 2025-07-17; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Toxicology; Bariatric Surgery Analgesia; Bariatric Surgery; Substance Use
Keywords: Metabolic bariatric surgery; toxicological screening; substance use; short-term outcomes; pain management; anesthesia requirements; postoperative complications; weight loss
MeSH Terms: conditions — Substance-Related Disorders; Agnosia; Postoperative Complications; Weight Loss | interventions — Urination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — clinical utility of routine preoperative toxicological screening tests (TST) in patients undergoing primary metabolic bariatric surgery (MBS). (Urine) All participants underwent comprehensive urine toxicological screening using a standardized multi-drug panel. The screening was performed using the Multi-Drug One Step Screen Test Panel (Urine) with reference number DOA-174, lot number 0000661863, with an expiry date of December 17, 2024. This dipstick test provided rapid, point-of-care screening for a comprehensive range of substances commonly encountered in clinical practice.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TST-positive: The toxicological panel tested for seven major categories of substances:
  1. COC (Cocaine): Detection of cocaine metabolites indicating recent cocaine use
  2. AMP (Amphetamines): Screening for amphetamine and methamphetamine compounds
  3. THC (Tetrahydrocannabinol): Detection of cannabis metabolites
  4. MOP (Morphine/Opiates): Screening for morphine, codeine, and related opiate compounds
  5. TRA (Tramadol): Specific detection of tramadol, a commonly prescribed analgesic in the region
  6. BAR (Barbiturates): Detection of barbiturate compounds
  7. BZO (Benzodiazepines): Screening for benzodiazepine medications
  Interventions: Diagnostic Test: Multi-Drug One Step Screen Test Panel (Urine)
- TST-negative: patients that tested negative in the dipstick test.
  Interventions: Diagnostic Test: Multi-Drug One Step Screen Test Panel (Urine)

INTERVENTIONS:
Diagnostic Test: Multi-Drug One Step Screen Test Panel (Urine) — Tested positive
  Groups: TST-positive
Diagnostic Test: Multi-Drug One Step Screen Test Panel (Urine) — tested negative
  Groups: TST-negative

SUMMARY:
Background: Preoperative substance use is a growing concern in patients undergoing metabolic bariatric surgery (MBS), but its impact on short-term outcomes remains debated. This study evaluated the association between preoperative toxicological screening test (TST) results and perioperative outcomes, including anesthesia requirements, postoperative recovery, complications, and one-year weight loss in patients undergoing MBS.

Key Points

1. Preoperative toxicological screening identifies a significant proportion (15.1%) of patients undergoing metabolic bariatric surgery with recent substance use that may not be disclosed through self-reporting.
2. Patients with positive toxicological screening tests require significantly higher anesthesia doses, experience more severe postoperative pain, and have higher rates of complications and readmissions within 30 days.
3. While short-term weight loss outcomes at one year show modest differences between toxicological screening test-positive and negative patients, the perioperative risk profile suggests the need for tailored management strategies for patients with recent substance use.

DETAILED DESCRIPTION:
The Middle East and North Africa (MENA) region has experienced a particularly rapid increase in obesity prevalence over recent decades, with some countries reporting rates exceeding 35% among adults. This trend is attributed to rapid urbanization, economic development, adoption of Western dietary patterns, and reduced physical activity. The high prevalence of obesity in the MENA region has created an urgent need for effective treatment strategies, including metabolic bariatric surgery (MBS).

MBS has established itself as the most effective long-term treatment for severe obesity, offering substantial and sustained weight loss along with resolution of obesity-related medical problems. The field has evolved significantly over the past decades, with procedures such as laparoscopic sleeve gastrectomy (LSG), Roux-en-Y gastric bypass (RYGB), and one-anastomosis gastric bypass (OAGB) becoming standard treatments for patients with severe obesity. These procedures not only achieve significant weight reduction but also provide remarkable improvements in type 2 diabetes, hypertension, dyslipidemia, and other obesity-related conditions.

The success of MBS depends on careful patient selection, thorough preoperative evaluation, and appropriate perioperative management. Substance use has become an important consideration among the factors influencing surgical outcomes. Substance use can affect wound healing and adherence to postoperative care protocols, potentially compromising surgical outcomes.

Managing anesthesia for obesity surgery in patients with substance abuse disorders presents a complex array of challenges. Obesity complicates airway management, alters pharmacokinetics and dynamics, demanding careful drug dosing and vigilant cardiopulmonary monitoring. Furthermore, chronic opioid users exhibit exaggerated pain, requiring dose modifications perioperatively but escalating risks of respiratory depression and postoperative hyperalgesia or withdrawal. Cocaine and amphetamine abuse increase the risks of arrhythmias, hypertension, myocardial ischemia, and unpredictable interactions with anesthetic agents. There is a necessity for multidisciplinary comprehensive perioperative optimization, including addiction consultation, careful substance withdrawal management, individualized anesthetic and surgical plans, multimodal analgesia, and extended postoperative monitoring for the possibility of respiratory complications and acute withdrawal symptoms.

A recent study by Chao et al. examined the association between toxicology positivity and outcomes in MBS patients in a retrospective review of 1,057 patients who underwent laparoscopic sleeve gastrectomy or Roux-en-Y gastric bypass. They found that 12.7% of patients had positive toxicology testing, with benzodiazepines (5.6%), opiates (3.5%), and cotinine (2.0%) being the most common substances detected. Their study did not find significant associations between toxicology positivity and preoperative length of time, 30-day complications, readmissions, or one-year weight loss.

In a cross-sectional study of elective surgery patients, Amin et al. found a strong positive correlation between toxicological screening drug detection and propofol induction dose, pain scores, and hospital stay. Similar findings were reported by Clavijo et al. in a prospective observational pilot study of patients undergoing spine surgery. They found inconsistencies between self-reporting and toxicological screening test results in 88% of patients, with significant correlations between polypharmacy and increased anesthesia requirements.

The MENA region provides unique challenges concerning substance use assessment owing to cultural, religious, and legal factors that may impact disclosure. Substance use is often stigmatized and criminalized in many MENA countries, potentially leading to underreporting during clinical evaluations. Epidemiological statistics show that drug usage patterns in the MENA region deviate from worldwide trends, with specific concerns about tramadol, cannabis, and prescription drugs. Tobacco usage remains prevalent throughout the area, with worries raised regarding the use of traditional medicines such as khat in certain regions. These drug use patterns have significant consequences for surgical patients because they may influence perioperative treatment, anesthetic requirements, and postoperative recovery. The stigmatization and underreporting of drug addiction in the MENA region highlights the importance of objective assessment methods, such as toxicological screening, to identify patients who may require modified perioperative management for patient safety and optimal care delivery.

The role of preoperative toxicological screening has been the subject of increasing research interest, particularly in procedures requiring careful perioperative management and in areas of uncertainty about patients' substance use disclosure. Despite the growing body of literature on this topic, there remains a gap in knowledge regarding the specific impact of preoperative substance use on outcomes following MBS, particularly in the MENA region, where substance use patterns and disclosure behaviors may differ from Western populations. This prospective observational study addressed this gap by evaluating the association between preoperative toxicological screening results and their impact on perioperative anesthetic management and short-term outcomes following MBS in Egypt.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (≥18 years) with obesity who were scheduled to undergo primary MBS, including laparoscopic sleeve gastrectomy (LSG), Roux-en-Y gastric bypass (RYGB), or one-anastomosis gastric bypass (OAGB)
* Patient selection followed the 2022 American Society for Metabolic and Bariatric Surgery (ASMBS) and International Federation for the Surgery of Obesity and Metabolic Disorders (IFSO) guidelines for MBS

Exclusion Criteria:

* previous bariatric or major abdominal surgery
* emergency procedures
* chronic pain syndromes
* severe psychiatric illness
* patient refusal that would impair informed consent or compliance with study protocols
* inability to complete follow-up assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 1,260 patients were enrolled in the study and underwent preoperative toxicological screening tests (TST). The study population had a mean age of 38.4 ± 9.7 years, with a predominance of female patients (72.3%). The mean preoperative BMI was 44.2 ± 6.8 kg/m². Laparoscopic sleeve gastrectomy (LSG) was the most common procedure (68.3%), followed by one-anastomosis gastric bypass (OAGB, 21.4%) and Roux-en-Y gastric bypass (RYGB, 10.3%).
  Of the 1,260 patients, 190 (15.1%) tested positive on preoperative TST for at least one substance. The most detected substances were tramadol (52.6% of positive tests), cannabis (28.4%), benzodiazepines (15.8%), opiates (10.5%), amphetamines (7.9%), barbiturates (5.3%), and cocaine (2.6%). Multiple substances were detected in 18.4% of TST-positive patients. Figure 1 illustrates the distribution of substances detected in the TST-positive group.
Sampling Method: Probability Sample
Enrollment: 1260 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
history of specific substance use and /or detected by toxicological screening | within 30 days post operative
  To determine the prevalence and patterns of substance use detected by preoperative toxicological screening tests (TST) in patients undergoing metabolic bariatric surgery (MBS) in the MENA region.
  Additional information regarding prescription status (prescribed versus self-prescribed) was obtained through structured patient interviews conducted by trained clinical staff for differentiation between legitimate medical use and recreational or non-prescribed substance use.
Anesthesia-related outcomes included dosages of induction agents (specifically propofol) and perioperative opioid consumption (intraoperative fentanyl dose and postoperative morphine consumption). | within 30 days post operative
  Recovery parameters were assessed, including recovery time (measured in minutes from extubation till meeting discharge criteria from the operative theatre (OR) to the post-anesthesia care unit (PACU)) and recovery status evaluated through Richmond Agitation-Sedation Scale (RASS). The RASS is a 10-point scale that ranges from -5 to +4, designed to evaluate a patient's level of alertness and agitation during recovery. Levels -1 to -5 denote 5 levels of sedation; levels +1 to +4 describe increasing levels of agitation. RASS level 0 is "alert and calm.
Pain assessment | within 30 days post operative
  was conducted using the Visual Analog Scale (VAS), measured multiple times during the first postoperative day: baseline, 1 hour, 6 hours, 12 hours, and 24 hours post-surgery. The VAS is a validated tool for pain assessment that consists of a 10-cm horizontal line with endpoints representing "no pain" (0) and "worst possible pain" (10). Patients were given 3 mg morphine if VAS scores reached ≥ 4. The time to first opioid request was also recorded as an indicator of pain onset and severity.

SECONDARY OUTCOMES:
postoperative recovery parameter | during the first 24 hours after surgery.
  Recovery time, between the 2 groups of patients during the first 24 hours after surgery.
  General anesthesia recovery time is measured by assessing a patient's return to pre-anesthetic function, encompassing various domains including consciousness, cognitive function, and physical capabilities, with common tools like the QoR-15 scale being used to quantify quality of recovery. While patients typically begin to wake within minutes and may go home within hours, full recovery can take up to 24 hours or longer for some aspects, depending on the individual and the surgery.
postoperative recovery parameter | during the first 24 hours after surgery
  Postoperative pain scores between the 2 groups of patients during the first 24 hours after surgery.
  Post-operative pain after general anesthesia is measured using the Visual Analog Scale (VAS), a 100mm line representing pain intensity. Acceptable pain levels post-surgery are generally considered to be mild to moderate, often defined as NRS scores of 4 or less, or VAS scores of 33 or less.
postoperative recovery parameter | during the first 24 hours after surgery.
  Analgesic requirements between the 2 groups of patients during the first 24 hours after surgery.
  Measuring analgesia requirements during general anesthesia involves continuous physiological monitoring and the use of specialized indices to assess pain and nociception in real-time, allowing for titration of analgesic medications to effect and minimizing both under- and over-dosing.
  Standard Physiological Monitoring:
  Essential for overall patient safety and can provide indirect clues about pain or stress. This includes:
  Electrocardiography (ECG): Monitors heart rate and rhythm. Pulse Oximetry (SpO2): Measures oxygen saturation. Blood Pressure Monitoring (NIBP): Assesses cardiovascular stability. Capnography: Measures carbon dioxide exhaled, indicating ventilation adequacy. Temperature Measurement: Detects changes like hypothermia or fever.
preoperative substance use affects short-term weight loss | 12 months postoperative
  To determine whether preoperative substance use affects short-term weight loss outcomes and associated medical problem resolution at one year following MBS. (in kilograms and BMI measured by weight in kilograms and height in meters)

CONTACTS AND LOCATIONS:
Locations (1):
- The surgical department of Medical Research Institute Hospital, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The analysis will be performed on a blinded dataset after completing the medical/scientific review. All protocol violations will be identified and resolved, and the dataset will be declared complete. All data will be collected in a data management system (Castor EDC, Amsterdam, The Netherlands; https://www.castoredc.com), handled according to Good Clinical Practice guidelines, Data Protection Directive certificate, and complied with Title 21 CFR Part 11. Furthermore, the data centers where all the research data will be stored are certified according to ISO27001, ISO9001, and Dutch NEN7510.
  Can be asked by the contact person
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: whole study period
Access Criteria: Ask contact person